CLINICAL TRIAL: NCT05792059
Title: DevElopMent of Clinical PATHwaYs to the Diagnosis of Heart Failure With Preserved Ejection Fraction (EMPATHY-HF)
Brief Title: DevElopMent of Clinical PATHwaYs to the Diagnosis of Heart Failure With Preserved Ejection Fraction
Acronym: EMPATHY-HF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Medical Research Center for Therapy and Preventive Medicine (Other Government)
Responsible Party: Sponsor
Other Study IDs: 01-02/23
Record Dates: First submitted 2023-03-17; First posted 2023-03-30 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Heart Failure With Preserved Ejection Fraction (HFpEF)

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with HFpEF
- patients without HFpEF

SUMMARY:
Prevalence of heart failure with preserved ejection fraction (HFpEF) continues to increase in the developed world, likely because of the increasing life expectancy and an increasing number of elderly patients.

Transthoracic echocardiography is essential for the diagnosis of HFpEF according to the current guidelines. The HFA-PEFF and H2FPEF diagnostic algorithms rely on clinical characteristics and echocardiography findings that indicate the presence of diastolic dysfunction.

These diagnostic algorithms are not applicable in remote areas where expert echocardiography cannot be performed due to the absence of modern ultrasound systems and lack of qualified specialists. Therefore, it is important to develop an algorithm to evaluate pre-test probability of HFpEF without echocardiographic markers, so it can be easily used in the primary outpatient care setting by any specialist.

The aim of this study is to find the associations between clinical and epidemiological characteristics and changes of intracardiac hemodynamics in patients with dyspnea and decreased exercise tolerance.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients complaining of shortness of breath, with two or more chronic non-communicable diseases (patients with comorbidities)

Exclusion Criteria:

* Morbid obesity;
* Any chronic diseases in the stage of exacerbation and / or decompensation;
* Systemic diseases, cancer;
* Cardiac arrhythmias: persistent atrial fibrillation or paroxysmal atrial fibrillation with frequent paroxysms;
* History of myocardial infarction, stroke, heart failure with reduced ejection fraction;
* Storage diseases, hypertrophic cardiomyopathy, concentric hypertrophy;
* Congenital and acquired heart defect;

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients complaining of shortness of breath, with two or more chronic non-communicable diseases (patients with comorbidities)
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-02-09 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
An increased of post-exercise E/e' ratio | during diastolic stress test (baseline)
An increased of post-exercise pulmonary artery systolic pressure (PASP) | during diastolic stress test (baseline)

CONTACTS AND LOCATIONS:
Locations (1):
- National Medical Research Center for Therapy and Preventive Medicine, Moscow, Russia